CLINICAL TRIAL: NCT00306891
Title: Open-label, Randomised, Phase 2 Study in Patients With Advanced Solid Tumours to Determine Effect of Food Upon Pharmacokinetics of a Single Oral Dose of Cediranib (AZD2171, Recentin™), Followed by an Assessment of the Safety & Tolerability of Fixed and Individualised Daily Dosing
Brief Title: Effect of Food Upon Pharmacokinetics of Single Oral Dose of Cediranib (AZD2171, Recentin™)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D8480C00021; 2005-003441-13
Record Dates: First submitted 2006-03-23; First posted 2006-03-27 (Estimated); Results first posted 2012-11-01 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Cancer
Keywords: Advanced solid tumours; Advanced cancer; tumor; tumour; RECENTIN
MeSH Terms: conditions — Neoplasms | interventions — cediranib

ARMS (4):
- Cediranib 45 mg Fed (Experimental): Part A: Cediranib 45 mg Fed State
  Interventions: Drug: Cediranib
- Cediranib 45 mg Fasted (Experimental): Part A: Cediranib 45 mg Fasted State
  Interventions: Drug: Cediranib
- Cediranib 45 mg Fixed Dose (Experimental): Part B: Cediranib 45 mg Fixed Dose
  Interventions: Drug: Cediranib
- Cediranib 30 - 90 mg Dose Escalation (Experimental): Part B: Cediranib 30 - 90 mg Dose Escalation
  Interventions: Drug: Cediranib 30 - 90 mg

INTERVENTIONS:
Drug: Cediranib — 45 mg oral dose
  Other Names: RECENTIN™
  Arms: Cediranib 45 mg Fasted; Cediranib 45 mg Fed; Cediranib 45 mg Fixed Dose
Drug: Cediranib 30 - 90 mg — oral tablet dose escalation
  Other Names: RECENTIN™
  Arms: Cediranib 30 - 90 mg Dose Escalation

SUMMARY:
The purpose of this study is to determine whether food has any effect on a single dose of Cediranib (AZD2171, Recentin™)followed by an assessment of the safety and tolerability of fixed daily dosing in comparison to varying dose levels on a patient-by-patient basis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of advanced solid tumour.
* Ability to eat a high fat breakfast

Exclusion Criteria:

* Poorly controlled high blood pressure.
* History of significant gastrointestinal problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-06; Primary Completion 2008-01 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AZD2171 Medical Science Director, MD, Study Director — AstraZeneca
Locations (4):
- United Kingdom (4):
  - Research Site, Glasgow
  - Research Site, Headington
  - Research Site, London
  - Research Site, Manchester

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a two part study.Part A had two arms, fed/fasted and fasted/fed. Part B had two arms, a fixed dose arm and a dose escalation arm.Patients(pts)in Part A were allowed to go in to Part B. Pts who chose not to go in to Part B discontinued the study.Additionally new pts were recruited to Part B. In Parts A/B, there was a total of 60 pts.
Pre-assignment Details: 60 patients were enrolled though only 45 patients were randomized to Part A and 47 to Part B.
  Completion of Part B means completed at least 16 weeks of treatment.
Groups:
- Cediranib 30 to 90 mg Dose Escalation: Part B: Cediranib Dose Escalation
Period: Part A
Arm/Group | Cediranib 45 mg Fed | Cediranib 45 mg Fasted | Cediranib 45 mg Fixed Dose | Cediranib 30 to 90 mg Dose Escalation
Started | 23 | 22 | 0 | 0
Completed | 18 | 16 | 0 | 0
Not Completed | 5 | 6 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0
Not completed — Condition under investigation worsened | 2 | 2 | 0 | 0
Not completed — Incorrect enrol/entry crit not fulfilled | 0 | 1 | 0 | 0
Not completed — Partial bowel obstruction | 1 | 0 | 0 | 0
Not completed — Reaccumul. of ascites following drainage | 0 | 1 | 0 | 0
Not completed — Suspicion of second malignancy | 0 | 1 | 0 | 0
Not completed — QTC interval outwith elig. criteria | 1 | 0 | 0 | 0
Period: Part B
Arm/Group | Cediranib 45 mg Fed | Cediranib 45 mg Fasted | Cediranib 45 mg Fixed Dose | Cediranib 30 to 90 mg Dose Escalation
Started | 0 | 0 | 16 (In Part B: Cediranib 45 mg Fixed Dose 4 new patients were randomized) | 31 (in Part B: Cediranib Dose Escalation 11 new patients were randomized.)
Completed | 0 | 0 | 5 | 14
Not Completed | 0 | 0 | 11 | 17
Not completed — Death | 0 | 0 | 1 | 2
Not completed — Adverse Event | 0 | 0 | 5 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 1
Not completed — Condition under investigation worsened | 0 | 0 | 2 | 8
Not completed — Development of study specific disc crit. | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cediranib 45 mg Fed | Cediranib 45 mg Fasted | Cediranib 45 mg Fixed Dose | Cediranib 30 to 90 mg Dose Escalation | Total
Number analyzed (Participants) | 23 | 22 | 16 | 31 | 92
Age Continuous [Mean (Standard Deviation); unit: Years] | 58.6 (10.6) | 51.2 (14.8) | 56.4 (13.1) | 56.0 (13.5) | 56.0 (13.0)
Sex/Gender, Customized [Number; unit: participants]
  Female, Part A | 10 | 10 | NA — Cediranib 45 mg Fixed dose arm existed only in Part B. | NA — Cediranib 30 to 90 mg Dose Escalation existed only in Part B. | 20
  Male, Part A | 13 | 12 | NA — Cediranib 45 mg Fixed dose arm existed only in Part B | NA — Cediranib 30 to 90 mg Dose Escalation existed only in Part B. | 25
  Female, Part B | NA — Cediranib 45 mg Fed/Fasted existed only in Part A. | NA — Cediranib 45 mg Fasted/Fed existed only in Part A. | 8 | 12 | 20
  Male, Part B | NA — Cediranib 45 mg Fed/Fasted only in Part A. | NA — Cediranib 45 mg Fasted/Fed existed only in Part A. | 8 | 19 | 27

OUTCOME MEASURES:

1. Primary Outcome: Part A: Area Under Plasma Concentration-time Curve (AUC)
Description: Area under plasma concentration-time curve from zero to infinity
Time Frame: Measurements were collected up to 168 hours (following single dosing).
Measure: Geometric Mean (Full Range); unit: ng*h/mL
Arm/Group | Cediranib 45 mg Fed | Cediranib 45 mg Fasted
Number analyzed (Participants) | 30 | 32
ng*h/mL | 1920 [778 to 5760] | 2392 [604 to 5730]

2. Primary Outcome: Part A: Maximum Plasma (Peak) Concentration (Cmax)
Description: Maximum plasma drug concentration
Time Frame: Measurements were collected up to 168 hours (following single dosing).
Measure: Geometric Mean (Full Range); unit: ng/mL
Groups:
- Arm 1 - Cediranib 45 mg Fed: Part A: Cediranib 45 mg Fed State
- Arm 2 - Cediranib 45 mg Fasted: Part A: Cediranib 45 mg Fasted State
Arm/Group | Arm 1 - Cediranib 45 mg Fed | Arm 2 - Cediranib 45 mg Fasted
Number analyzed (Participants) | 31 | 33
ng/mL | 87.02 [27.6 to 265] | 127.9 [35.6 to 334]

3. Secondary Outcome: Part A: AUC (0-t)
Description: Area under the curve from time 0 to the last measureable time point
Time Frame: Measurements were collected up to 168 hours (following single dosing).
Measure: Geometric Mean (Full Range); unit: ng*h/mL
Arm/Group | Arm 1 - Cediranib 45 mg Fed | Arm 2 - Cediranib 45 mg Fasted
Number analyzed (Participants) | 30 | 32
ng*h/mL | 1896 [764 to 5700] | 2348 [599 to 5290]

4. Secondary Outcome: Part A: Time to Peak or Maximum Concentration (Tmax)
Description: Time to reach peak or maximum concentration or maximum response
Time Frame: Measurements were collected up to 168 hours (following single dosing).
Measure: Geometric Mean (Full Range); unit: hr
Arm/Group | Arm 1 - Cediranib 45 mg Fed | Arm 2 - Cediranib 45 mg Fasted
Number analyzed (Participants) | 31 | 33
hr | 4.59 [2.0 to 25] | 3.52 [2.0 to 6.1]

5. Secondary Outcome: Part A: Terminal Phase Half-life (t1/2λz)
Description: Terminal phase half-life
Time Frame: Measurements were collected up to 168 hours (following single dosing).
Measure: Geometric Mean (Full Range); unit: hr
Arm/Group | Arm 1 - Cediranib 45 mg Fed | Arm 2 - Cediranib 45 mg Fasted
Number analyzed (Participants) | 30 | 32
hr | 23.99 [12.1 to 37.5] | 24.72 [10.2 to 60.2]

6. Secondary Outcome: Part A: Apparent Total Body Clearance (CL/F)
Description: Apparent total body clearance of drug from plasma
Time Frame: Measurements were collected up to 168 hours (following single dosing).
Measure: Geometric Mean (Full Range); unit: L/h
Arm/Group | Arm 1 - Cediranib 45 mg Fed | Arm 2 - Cediranib 45 mg Fasted
Number analyzed (Participants) | 30 | 32
L/h | 23.44 [7.81 to 57.8] | 18.81 [7.85 to 74.5]

7. Secondary Outcome: Part B: Best Overall Response Rate (ORR)
Description: Evaluation of target lesions Complete Response(CR)Disappearance of all target lesions Partial Response(PR) At least a 30% decrease in the sum of LD(longest diameter)of target lesions taking as reference the baseline sum LD.Progressive Disease(PD).At least a 20% increase in the sum of LD of target lesions taking as references the smallest sum LD recorded(either at baseline or at previous assessment since treatment began).Stable Disease(SD) Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.Note: Appearance of new lesions only counts towards the overall visit response,not towards the response of target or non-target lesions.
  Evaluation of non-target lesions Complete Response(CR)Disappearance of all non-target lesions Non-Complete Response(non-CR/Non-Progression[non-PD])Persistence of one or more non-target lesion or/and maintenance of tumour marker level above the normal limits.Progression(PD)Unequivocal progression of existing non-target lesions
Time Frame: Baseline, week 8, week 16 and every 8 weeks thereafter until discontinuation.
Population: ITT (intention-to-treat ) patients with baseline RECIST data
Measure: Number; unit: Participants
Groups:
- Arm 3 - Cediranib 45 mg Fixed Dose: Part B: Cediranib 45 mg Fixed Dose
- Arm 4 - Cediranib 30-90 mg Dose Escalation: Part B: Cediranib 30-90 mg Dose Escalation
Arm/Group | Arm 3 - Cediranib 45 mg Fixed Dose | Arm 4 - Cediranib 30-90 mg Dose Escalation
Number analyzed (Participants) | 15 | 29
Participants | 1 | 3

8. Secondary Outcome: Part B: Progression-free Survival (PFS)
Description: Target lesions: Progressive Disease (PD) At least a 20% increase in the sum of LD (longest diameter)of target lesions taking as references the smallest sum LD recorded (either at baseline or at previous assessment since treatment began).
  Non target lesions: Persistence of one or more non-target lesion or/and maintenance of tumour marker level above the normal limits.
  Progression (PD) Unequivocal progression of existing non-target lesions.
Time Frame: Number of days from randomisation until progressive disease based on RECIST (progression of target lesions, clear progression of existing non-target lesions or the appearance of one or more new lesions) or death in the absence of progression.
Population: ITT (intention-to-treat ) patients with baseline RECIST data.One patient was randomized and had baseline RECIST assessments, but did not have any further RECIST assessments. Therefore they were censored at baseline, meaning the lowest value in the range was set to zero.
Measure: Median (Full Range); unit: Days
Arm/Group | Arm 3 - Cediranib 45 mg Fixed Dose | Arm 4 - Cediranib 30-90 mg Dose Escalation
Number analyzed (Participants) | 15 | 29
Days | 135 [39 to 314] | 139 [0 to 454]

ADVERSE EVENTS:
Groups:
- Cediranib 45 mg Part A: Part A: Cediranib 45 mg
- Cediranib 30 - 90 mg Dose Escalation: Cediranib 30 - 90 mg Dose Escalation
Arm/Group | Cediranib 45 mg Part A | Cediranib 45 mg Fixed Dose | Cediranib 30 - 90 mg Dose Escalation
Serious Adverse Events (participants affected / at risk) | 6/39 | 9/16 | 20/31
Other Adverse Events (participants affected / at risk) | 34/39 | 16/16 | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cediranib 45 mg Part A (N=39) | Cediranib 45 mg Fixed Dose (N=16) | Cediranib 30 - 90 mg Dose Escalation (N=31)
Angina Pectoris (Cardiac disorders) | 1 | 1 | 0
Cardiac Failure (Cardiac disorders) | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 3
Vomiting (Gastrointestinal disorders) | 0 | 0 | 3
Abdominal Pain Lower (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 0 | 1
Gastric Perforation (Gastrointestinal disorders) | 0 | 1 | 0
Gastric Ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal Perforation (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal Perforation (Gastrointestinal disorders) | 0 | 1 | 0
Large Intestine Perforation (Gastrointestinal disorders) | 0 | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 1
Bile Duct Obstruction (Hepatobiliary disorders) | 0 | 0 | 1
Jaundice Cholestatic (Hepatobiliary disorders) | 0 | 1 | 0
Central Line Infection (Infections and infestations) | 0 | 0 | 1
Clostridial Infection (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 0
Viral Labyrinthitis (Infections and infestations) | 1 | 0 | 0
Tracheostomy Malfunction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intracranial Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Spinal Cord Compression (Nervous system disorders) | 0 | 0 | 1
Suicide Attempt (Psychiatric disorders) | 0 | 0 | 1
Renal Disorder (Renal and urinary disorders) | 1 | 0 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 0 | 1
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cediranib 45 mg Part A (N=39) | Cediranib 45 mg Fixed Dose (N=16) | Cediranib 30 - 90 mg Dose Escalation (N=31)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 3
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 1
Haemoglobinaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 1
Bradycardia (Cardiac disorders) | 2 | 0 | 1
Bundle Branch Block Right (Cardiac disorders) | 0 | 1 | 0
Deafness Unilateral (Ear and labyrinth disorders) | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 4
Dry Eye (Eye disorders) | 0 | 2 | 0
Visual Disturbance (Eye disorders) | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 5 | 13 | 25
Nausea (Gastrointestinal disorders) | 9 | 11 | 17
Vomiting (Gastrointestinal disorders) | 4 | 10 | 14
Constipation (Gastrointestinal disorders) | 4 | 10 | 10
Abdominal Pain (Gastrointestinal disorders) | 1 | 4 | 9
Stomatitis (Gastrointestinal disorders) | 0 | 4 | 9
Dry Mouth (Gastrointestinal disorders) | 1 | 1 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 3 | 3
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 1 | 1
Epigastric Discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Lip Blister (Gastrointestinal disorders) | 0 | 1 | 0
Mouth Ulceration (Gastrointestinal disorders) | 0 | 1 | 0
Oral Pain (Gastrointestinal disorders) | 0 | 1 | 1
Tongue Ulceration (Gastrointestinal disorders) | 0 | 1 | 0
Fatigue (General disorders) | 8 | 5 | 10
Oedema Peripheral (General disorders) | 2 | 1 | 4
Pyrexia (General disorders) | 0 | 0 | 2
Unevaluable Event (General disorders) | 0 | 0 | 2
Malaise (General disorders) | 0 | 1 | 0
Oral Candidiasis (Infections and infestations) | 1 | 1 | 3
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 2
Rhinitis (Infections and infestations) | 0 | 2 | 1
Tooth Abscess (Infections and infestations) | 0 | 2 | 1
Neutropenic Sepsis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Postoperative Wound Infection (Infections and infestations) | 0 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 1
Vaginal Candidiasis (Infections and infestations) | 0 | 1 | 1
Viral Infection (Infections and infestations) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 2
Weight Decreased (Investigations) | 1 | 2 | 8
Blood Thyroid Stimulating Hormone Increased (Investigations) | 0 | 2 | 7
Alanine Aminotransferase Increased (Investigations) | 0 | 1 | 2
Blood Pressure Increased (Investigations) | 2 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 0 | 1 | 1
Liver Function Test Abnormal (Investigations) | 0 | 1 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 4 | 8
Anorexia (Metabolism and nutrition disorders) | 3 | 3 | 6
Alkalosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Metabolic Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 4
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Mobility Decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Lethargy (Nervous system disorders) | 8 | 4 | 7
Dizziness (Nervous system disorders) | 2 | 1 | 6
Headache (Nervous system disorders) | 2 | 5 | 5
Dysgeusia (Nervous system disorders) | 0 | 1 | 1
Neuralgia (Nervous system disorders) | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 3
Anxiety (Psychiatric disorders) | 2 | 1 | 0
Depressed Mood (Psychiatric disorders) | 2 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 2
Urinary Tract Disorder (Renal and urinary disorders) | 0 | 1 | 0
Urine Odour Abnormal (Renal and urinary disorders) | 0 | 1 | 0
Amenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 3 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Skin Induration (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 9 | 10 | 23
Hypotension (Vascular disorders) | 0 | 1 | 0
Lymphoedema (Vascular disorders) | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a Study Site or an Investigator requests permission to publish data from this study, any such publication (including oral presentations) is to be agreed with AstraZeneca prior to publication.